CLINICAL TRIAL: NCT05605301
Title: Pharmacokinetics Study of Oral 2-Deoxy-D-Glucose (2DG) in Subjects With a Confirmed Diagnosis of Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Epilepsy Foundation (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Nathan Fountain, MD, Professor of Epileptology and Neurology, University of Virginia
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSR210085
Record Dates: First submitted 2022-10-22; First posted 2022-11-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy | interventions — Deoxyglucose

STUDY DESIGN:
Intervention Model Description: Subjects will be given 2DG orally during a single day of dosing at one of three sequential dose levels (a single dose of 40 mg for Dose Level 1, a single dose of 60 mg for Dose Level 2, or 60 mg bid for Dose Level 3). The total dose will not exceed 120 mg/day, or 60 mg maximum.
  as a single dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential ascending dose cohort (Experimental): Cohort 1 will receive single 40 mg dose once. Cohort 2 will receive single 60 mg dose once. Cohort 3 will receive (2) 60 mg dose on one occasion.
  Interventions: Drug: Oral 2-Deoxy-D-Glucose (2DG)

INTERVENTIONS:
Drug: Oral 2-Deoxy-D-Glucose (2DG) — 2DG will be formulated as an solid dosage form and administered orally.

SUMMARY:
This project studies how 2-deoxy-glucose (2DG) pills are absorbed and distributed in people with epilepsy. 2DG is similar to glucose, the main energy source for the brain, but it cannot be used as energy. During seizures, neurons are at a very high metabolic state with huge glucose metabolism as glycolysis is accelerated to supply the high metabolic needs of a seizure. 2DG is taken up by cells but cannot be metabolized by the first enzyme in the glycolytic pathway, thus is stops, or "clogs up", glycolysis. Since brain metabolism is almost entirely dependent on glucose as an energy source, glycolysis is arrested and may stop seizures. It is hoped that 2DG will stop seizures by interfering with the brain's energy use.

This is an open-label phase 2 study of the pharmacokinetics (PK), safety, and tolerability of 2DG administered orally to adult epilepsy patients. A 3-level 2DG dose escalation is planned in sequential cohorts of 3 subjects in each cohort with review of each cohort before proceeding to the next cohort. On the day of oral 2DG exposure, subjects will receive a single dose of 40 mg in the first cohort, a single dose of 60 mg in the second cohort, and two 60 mg doses (60 mg bid) in the third cohort.

After 3 subjects have completed dosing at Dose Level 1 (40 mg/day), the safety and PK results will be reviewed. The Study Committee will determine if the next cohort should be enrolled at Dose Level 2 (60 mg/day). The same procedure will be repeated to determine if the next cohort should be enrolled at Dose Level 3 (60 mg bid = 120 mg/day). If the Study Committee determines that the most recent dose is not tolerated or that there are significant adverse events, the subsequent Dose Level will not be enrolled.

A standard time-concentration curve will be constructed from the 2DG levels obtained from the PK blood draws. Parameters will be calculated for: time to maximum concentration (tmax), maximum concentration (Cmax), elimination rate, half-life (t1/2), AUC, and derived parameters. Statistical analysis will not be performed because of the small n, but this will nevertheless establish the PK profile of 2DG in people with epilepsy. The most important parameter will be the AUC which determines drug exposure.

DETAILED DESCRIPTION:
The study will be conducted as a 1-day Monitored Dosing and Pharmacokinetics Period in an inpatient setting. Subjects will report to the hospital in a fasted state (since midnight) on the morning of the pharmacokinetics study. Subjects will continue to fast until one hour after the 2DG dose has been given. 2DG will be given as either a single oral dose (40 mg for Dose Level 1; 60 mg for dose level 2) or 60 mg bid (Dose Level 3). Blood for pharmacokinetic analysis will be drawn at time 0 (prior to drug administration), and then at 15, 30, 45, and 60 minutes and at 2, 4, 6, 12, and 24 hours after single dose 2DG administration. Blood for pharmacokinetic analysis will be drawn at time 0 (prior to drug administration) and then at 15, 30, 45, and 60 minutes and at 2, 4, 6, 12, and 24 hours after the last dose for Dose Level 3. Patients will be closely monitored for safety during and following dosing with 2DG.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of epilepsy. For the purpose of inclusion, the seizure types include complex partial, simple partial motor, primary generalized tonic-clonic, secondary generalized tonic-clonic, tonic, clonic and atonic seizures, as well as simple partial and absence seizures.

  * Stable treatment regimen with no change in antiepileptic drugs or antiepileptic drug doses for 28 days prior to enrollment.
  * Women of childbearing potential must be using a standard method of birth control and agree not to become pregnant during the trial. Men must agree to not father a child during the trial.
  * BMI must be between 18 and 35.

Exclusion Criteria:

* Occurrence of non-epileptic psychogenic spells within 2 years prior to enrollment.
* Current or past history of diabetes or any abnormality of glucose metabolism.
* Use of glucocorticoids, hypoglycemic agents (e.g. metformin) or any drug that alters glucose levels.
* Use of any drug that is expected to alter glucose absorption, metabolism or serum measurements.
* Clinically significant psychiatric or medical disease.
* Previous therapeutic use of 2DG.
* Pregnant or nursing women.
* Use of an investigational medication within 2 months prior to enrollment.
* Supine systolic blood pressure < 90 or > 160 mm Hg or diastolic > 90 mm Hg, or pulse < 60 or > 110 BPM.
* Clinically significant abnormal 12-lead ECG.
* Baseline prolongation of the QTc interval > 450 msec.
* Clinically significant abnormal result by speckle tracking echocardiography (STE).
* Elevated ALT or AST more than 1.5 times upper reference limit.
* Baseline fasting glucose < 60 or > 110.
* History of status epilepticus within 6 months prior to enrollment.
* Progressive structural brain lesion or illness likely to progress during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Collected from time of drug administration to 24 hours post dose
  AUC will be calculated from 2DG blood levels collected at time 0, 15, 30, 45, and 60 minutes and at 2, 4, 6, 12, and 24 hours after single dose of 2DG.
Incidence of Treatment-Emergent Adverse Events | From time of drug administration until 24 hours post-dose
  Spontaneously reported adverse events will be summarized by type and severity by the most recent version of MedRA terminology. Adverse events will be graded as mild, moderate, or severe and by whether the relationship to study drug is related, possibly related, or unrelated.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan B Fountain, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No